CLINICAL TRIAL: NCT04244669
Title: The Impact of Different Spinal Cord Stimulation Waveforms on Quality of Life in Patients With Chronic Pain (SCS-Quality)
Brief Title: Impact of the SCS With Different Waveforms Over the Quality of Life (SCS-Quality)
Acronym: SCS-Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pablo López Pais (Other)
Responsible Party: Sponsor-Investigator, Pablo López Pais, Principal Investigator, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCS-Quality
Record Dates: First submitted 2019-11-24; First posted 2020-01-28 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Failed Back Surgery Syndrome; Spinal Cord Stimulation
Keywords: FBSS; SCS; HD; Quality of life; Pain; Activity monitoring
MeSH Terms: conditions — Failed Back Surgery Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multicentre, parallel, controlled, and double-blind trial. It is a study with 2 groups with evaluation pre and post treatment with SCS implantation. The study has been designed to assess primarily non-inferiority and secondarily superiority of SCS DTM therapy
Who Masked: Care Provider, Investigator
Masking Description: The patient will not informed about the treatment arm, but the presence of paresthesia is a factor that break the masking.
  The care provider and investigators will not know the treatment arm and only collect the information in the forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SCS with Conventional Stimulation (Experimental): In this group, a conventional stimulation with low frequency will be tried. It will be programmed according to the usual clinical practice looking for one or more combinations of poles that allow a coverage of paraesthesia with a conventional stimulation of at least 80% of the painful area. This programming will be modified until getting not only 80% coverage but also a decrease of at least 50% of pain in that area.
  Interventions: Device: IPG with Conventional Stimulation
- SCS with SCS DTM Stimulation (Experimental): IIn this group the SCS DTM™ workflow will be programmed. Each SCS DTM™ program group has at least two programs with different pulse rate in the 20 to 1,200 Hz range and each having a maximum pulse width of 1ms.
  Interventions: Device: IPG with SCS DTM

INTERVENTIONS:
Device: IPG with Conventional Stimulation — In this group, a conventional stimulation with low frequency will be tried. It will be programmed according to the usual clinical practice looking for one or more combinations of poles that allow a coverage of paraesthesia with a conventional stimulation of at least 80% of the painful area. This programming will be modified until getting not only 80% coverage but also a decrease of at least 50% in that area. It can be reprogrammed as many times as necessary during the 14-21 days of margin.
  Arms: SCS with Conventional Stimulation
Device: IPG with SCS DTM — In this group the SCS DTM™ workflow will be programmed. Each SCS DTM™ program group has at least two programs with different pulse rate in the 20 to 1,200 Hz range and each having a maximum pulse width of 1ms
  Arms: SCS with SCS DTM Stimulation

SUMMARY:
Prospective, randomized, multicentre, parallel, controlled, and double-blind trial. It is a study with 2 groups with evaluation pre and post treatment with Spinal Cord Stimulation (SCS) implantation of patients with Failed Back Surgery Syndrome (FBSS). The study has been designed to assess primarily non-inferiority and secondarily superiority of SCS DTM therapy

DETAILED DESCRIPTION:
Over 18 years old patients, with leg with or without low back neuropathic pain (DN4 ≥4), previously undergoing low back surgery that, after an Evidence-Based (EB) medical therapy, can be eligible to SCS therapy following the Good Clinical Practice (GCP) guidelines will be implanted of two leads in the epidural thoracic level with at least two poles (Medtronic Vectris) covering the T9-T10 interspace and, if the trial is positive, a Medtronic Intellis Internal Pulse Generators (IPG) will be implanted.

The patients will be randomized to two groups to compare the improvement of pain control, the functional state and the quality of life of the patients by SCS Therapy across 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Leg with/without Low back pain with neuropathic characteristics (VAS ≥ 5 and DN4≥4) during at least 6 months before the screening consultation.
* Stable medical therapy with Evidence Based Medicine (EBM) during at least one month before the screening
* Ready and able to accomplish the procedures of the study and use the activity monitor and the medication diary.
* Have 18 years old or older when the patient signs the informed consent
* Pain kept during at least the last 6 months with VAS ≥ 6 and functional limitation due to the pain
* Refractory to treatment (during at least 3 months), and/or
* Intolerable adverse effects that avoid an optimum medical treatment
* Previous lumbosacral surgery for treatment of the cause of his pain
* Pain attributable to a low back pathology

Exclusion Criteria:

* Pregnant or with planned pregnancy
* Life expectancy <1 year.
* Polyneuropathy.
* Important Heart disease or peripheral vascular disease
* Degenerative disease that can decrease the functional capacity
* Alcoholism - Drug abuse
* Active infection
* Oncological active disease
* Haematological disorder with increased bleeding risk
* Patient unable to understand / follow the target of the study and the work flow
* When trial period has finished, the negative clinical response will be considered an exclusion criterion. The treatment could be completed, and the data collected but the patient will be excluded of the Randomized Clinical Trial (RCT) and the data analysed separately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority VAS | 3, 6,12 months
  Non-inferiority of SCS DTM therapy compared with low frequency SCS in change of quantitative measure of pain with Visual Analogue Scale (VAS, 0-10 points, no pain to the worst pain imaginable).

SECONDARY OUTCOMES:
Superiority VAS | 3, 6,12 months
  Superiority of SCS DTM therapy compared with low frequency SCS in the quantitative measure of pain with Visual Analogue Scale (VAS, 0-10, no pain to the worst pain imaginable).
Correlation between VAS and functionality and quality of life scores | 3, 6,12 months
  Correlation between the change of Visual Analogue Scale (VAS, 0-10, from no pain to the worst pain imaginable) and functionality (Oswestry Disability Index, ODI, from 0 to 100% of disability due to low back pain; Short form 36, SF-36, 0-100 points, from the worst health to the better) and quality of life scores (EuroQol-5D, EQ-5D, 0-1, from death to the best state of health)
Objective measure of activity parameters | 3, 6,12 months
  Difference between SCS DTM therapy compared with low frequency SCS in Objective measure of activity parameters (measured with an activity monitor)
Qualitative measure of dream quality | 3, 6,12 months
  Qualitative measure of dream quality Pittsburgh Sleep Quality Index (PSQI, 0 to 21, where lower scores denote a healthier sleep quality)
Scores/Questionnaires of disability: ODI | 3, 6,12 months
  Differences in Oswestry Disability Index versus control and between the arms (ODI, from 0 to 100% of disability due to low back pain)
Scores/Questionnaires of quality of life: SF-36 | 3, 6,12 months
  Differences in Short Form 36 versus control and between the arms (SF-36, 0-100 points, from the worst health to the better)
Scores/Questionnaires of quality of life: EQ-5D | 3, 6,12 months
  Differences in EQ-5D versus control and between the arms (EuroQol-5D, EQ-5D, 0-1, from death to the best state of health)
Medication consumption | 3, 6,12 months
  Medication consumption changes measured with Medication Quantification Scale III (MQSIII, from 0 points, no medication, according to the doses of each analgesic drug applying adjustment factors)
Observational parameters: ratio of adverse effects | 3, 6,12 months
  Observational parameters: ratio of adverse effects
Observational parameters: time of battery charge | 3, 6,12 months
  Observational parameters: time of battery charge
Observational parameters: quality of battery charge | 3, 6,12 months
  Observational parameters: quality of the battery recharge measured with the parameter provided by the IPG (Internal Pulse Generator), which classifies as bad, good or excellent
Changes in quality of life assessed by wrist activity monitor accelerometer | 3, 6,12 months
  To develop activity parameters measurables with an activity monitor and applicable clinically applying big data and complex mathematical calculations of position vectors and gyroscope data and activity monitor accelerometer, to predict changes early
Changes in VAS assessed by wrist activity monitor accelerometer | 3, 6,12 months
  To develop activity parameters measurables with an activity monitor and applicable clinically applying big data and complex mathematical calculations of position vectors and gyroscope data and activity monitor accelerometer, to predict changes early

CONTACTS AND LOCATIONS:
Locations (1):
- Pablo López Pais, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No